CLINICAL TRIAL: NCT05407012
Title: TRANS-FOODS: Preventing Peanut Allergy Through Improved Understanding of the Transcutaneous Sensitisation Route, Novel Food Processing and Skin Care Adaptations
Acronym: TRANS-FOODS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: University Hospital, Bonn (Other); Institut Curie (Other); Charite University, Berlin, Germany (Other); Levantine UK (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RE19787
Record Dates: First submitted 2022-05-26; First posted 2022-06-07 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Allergy;Food; Food Allergy Peanut; Pathways and Sources of Exposure
Keywords: Allergy; Food safety; Public health; Dermatology; Food manufacture
MeSH Terms: conditions — Food Hypersensitivity; Peanut Hypersensitivity; Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention of the barrier enhancing preparation (Experimental): Dry skin or atopic dermatitis or healthy skin; application of the peanut protein extract +/- massage after extract application.
  Interventions: Other: Application of the barrier enhancing preparation.
- Absence of the barrier enhancing preparation (No Intervention): Dry skin or atopic dermatitis or healthy skin; application of the peanut protein extract +/- massage after extract application.

INTERVENTIONS:
Other: Application of the barrier enhancing preparation. — Application of the barrier enhancing preparation around 30 minutes before application of the peanut protein extract +/- massage after extract application;
  Arms: Intervention of the barrier enhancing preparation

SUMMARY:
This project aims to study the immune responses to peanut allergen in those with a skin barrier defect with and without skin massage, specifically it aims to:

1. Establish if peanut allergen components can pass into human skin through regular massage using the peanut protein-containing extract.
2. Clarify whether this effect is amplified in those with an impaired skin barrier (AD and dry skin vs healthy controls).
3. Assess whether peanut protein components can be detected in interstitial skin fluid (ISF) using a suction device.
4. Test whether peanut protein components present in ISF are able to induce activation of basophils in blood of peanut allergic donors.
5. Assess whether the transcutaneous uptake of peanut protein can be reduced by the prior use of a barrier enhancing cream.

DETAILED DESCRIPTION:
The study aims to understand how peanut processing methods and peanut co-administration with oils, as is standard during the industrial processing of peanuts, influences the development of peanut allergy through the skin.

Cutaneous exposure of allergens is a crucial, but hitherto under explored route of food sensitisation, that if understood could lead to the development of translatable strategies to prevent food allergy. Food processors require a greater understanding of how allergen exposure cause allergy so that they can adapt their processing methods to counteract these exposure processes. Furthermore, this proposed research aligns with on-going efforts across Europe to address the increasing problems associated with food allergy but it is unique in that it focuses on cutaneous allergen exposure, which is a field in desperate need of more systematic study.

The assembled team of investigators (from the UK, Germany and France) joined by a peanut industry partner (Levantine) and patient and consumer representatives will aim to address the following hypotheses:

Understanding the mechanisms by which:

* Peanut proteins pass into the skin via the appendages to trigger an immune response.
* Skin stretching that occurs during massage opens up the skin appendages allowing more peanut protein into the skin and leads to dendritic cell activation and induction of T helper 2 cell response.
* Co-administration of peanut proteins and an oil to the skin increases allergenicity.
* Skin barrier impairment and inflammation (AD) increases allergenicity.

Test novel approaches to peanut allergy prevention whereby:

* Modifications in peanut processing can reduce allergen exposure via the skin.
* Meticulous hand hygiene reduces skin contamination with peanut protein.
* Application of a barrier enhancing cream can strengthen the skin barrier, in particular in those with atopic dermatitis, and reduce the risk of transcutaneous sensitisation further.

ELIGIBILITY:
Inclusion Criteria:

* Adult healthy volunteers (50% of the cohort), and adults with dry skin and AD (fulfilling the refined Hanifin and Rajka criteria, 50% of the cohort).
* Willingness to apply the study intervention and to not use any other topical preparations over theforearms during the study period.

Exclusion Criteria:

* History of peanut allergy.
* Positive skin prick test to peanut (>0 mm).
* No regular consumption of peanut products.
* Widespread AD, in particular if this involves the test sites of the forearms.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-04-05 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Detection of peanut protein components (μg of the proteins per cm² of skin) in retrieved interstitial fluid. | 8 weeks
  Detection of peanut protein components (μg of the proteins per cm² of skin) in retrieved interstitial fluid.
Activation of blood basophil from peanut allergic donors (measured as %CD63-positive basophils) by peanut proteins present in interstitial fluid. | 8 weeks
  Activation of blood basophil from peanut allergic donors (measured as %CD63-positive basophils) by peanut proteins present in interstitial fluid.

SECONDARY OUTCOMES:
Detection of inflammatory cytokine markers (IL-4, IL-13, IL-33 and TSLP) in interstitial fluid. | 8 weeks
  Detection of inflammatory cytokine markers (IL-4, IL-13, IL-33 and TSLP) in interstitial fluid.
Raised transepidermal water loss. | 8 weeks
  Raised transepidermal water loss.

OTHER OUTCOMES:
Assess skin barrier function measures (skin surface pH). | 8 weeks
  Assess skin barrier function measures (skin surface pH).

CONTACTS AND LOCATIONS:
Overall Officials: Carsten Flohr, Principal Investigator — King's College London
Locations (1):
- Unit for Population-Based Dermatology Research, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No